CLINICAL TRIAL: NCT06891768
Title: Bacteriological Profile and Antibiotic Sensitivity in Neonatal Intensive Care Unit At Assuit University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madleen Thabet Hofni Basali, Doctor, Assiut University
Other Study IDs: Ab sensitivity in neonates
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Nosocomial Infection in Neonatal Intensive Care Unit
MeSH Terms: interventions — Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Blood culture — Blood culture for bacteriological profile and antibiotic sensitivity

SUMMARY:
The study aims to assess the bacteriological profile and antibiotic sensitivity in NICU of pediatric hospital of assuit university.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines nosocomial infections (NI), also referred to as healthcare-associated infections (HAI's), as illnesses that develop in a patient while they are receiving treatment in a hospital or other healthcare institution but were neither present nor incubating at the time of admission . The symptoms should appear at least 2 calendar days admission to the hospital . The severity of the illness, prematurity, congenital defects, systemic diseases, degree of invasive monitoring, indiscriminate use of antibiotics, failures in sterilisation and disinfection techniques, and the type of diagnostic procedures all directly increase the risk of nosocomial infection in neonates . Long hospital stays, permanent incapacity, heightened antibiotic resistance in microorganisms, significant additional expenses for health systems, high costs for patients and their families, and avoidable deaths are all consequences of nosocomial infections . The most commonly encountered HAI's are central line associated blood stream infection (CLABSI), ventilator associated pneumonia (VAP), catheter associated urinary tract infection (CAUTI) and surgical site infections (SSI's). The other possible HAI's include meningitis, conjunctivitis and skin infections . The symptoms of health-associated infections are typically nonspecific and resemble those of other frequent neonatal diseases, including metabolic, respiratory, and thermoregulatory problems.However, improving an infant's prognosis requires prompt care. Typically, antimicrobial treatment is started without laboratory verification . Annually, more than a million neonatal deaths occur globally, with 30%-40% of these fatalities in low-resource nations linked to infections acquired in hospitals. In the NICU, bacteria, fungi, and viruses can persist and contaminate surfaces, equipment, and the surrounding environment for different lengths of time . In assuit university there is a study that has done about the incidence and risk factors of health care associated infections in NICU and it stated that out of 150 neonates , 107 developed nosocomial infection ,As regards the microbial profile and the distribution of isolated microorganisms from positive blood cultures, the most common pathogens were Staphylococcus aureus (22.7%) .The most common isolated microorganisms from positive endotracheal aspirate cultures were Klebsiella spp. (16%) . A study from Cairo university included 153 cases of neonatal sepsis; 63 (41.2%) EOS and 90 (58.8%) LOS. The majority of the neonates had very low or moderately low birth weight (90.9%). All neonates received first-line antibiotics in the form of ampicillin-sulbactam, and gentamicin. Second-line antibiotics were administered to 133 neonates (86.9%) as vancomycin and imipenem-cilastatin. Mortalities were more common among EOS group (p < 0.017). Positive blood cultures were detected in 61 neonates (39.8%) with a total number of 66 cultures. The most commonly encountered organisms were Klebsiella MDR and CoNS (31.8% each). Klebsiella MDR was the most predominant organism in EOS (28.9%), while CoNS was the most predominant in LOS (39.2%) The detected organisms were divided into 3 families; Enterobacteriaceae, non-fermenters, and Gram-positive family. There 3 families were 100% resistant to ampicillin. The highest sensitivity in Enterobacteriaceae and Non-fermenters was for colistin and polymyxin-B. An HSS of 3-8 had a sensitivity and specificity of 62.3% and 57.6%, respectively for diagnosis of culture-proven sepsis . A study from Ain Shams university included a 1-year records of a total of 1280 pathogens were studied. The highest number of pathogens were isolated from blood cultures (44.84%), followed by urine (41.41%) then wound swabs (13.75%). Gram-negative isolates (57.5%) were more prevalent than gram-positive ones (31.1%). The most frequently isolated pathogens were Klebsiella spp. (22.5%), Escherichia coli (13.4%), and Coagulase-negative Staphylococci (12.5%). The highest percentage of resistance among gram-positive organisms was exhibited by penicillin (89.5%) followed by erythromycin (83.98%) and then cefoxitin (76.52%). None of the isolates showed resistance to linezolid and resistance to vancomycin was minimal (2.62%). Gram-negative isolates exhibited high overall resistance to all used antibiotic classes. The least frequency of resistance was recorded against nitrofurantoin (52.5%), amikacin (58.01%), followed by imipenem (59.78%) and meropenem (61.82%). All isolates of Pseudomonas and Acinetobacter showed 100% susceptibility to colistin . Therefore, this study was done to know the bacteriological profile and the culture sensitivity of nosocomial infection in neonatal intensive care unit in pediatric hospital of assuit university.

ELIGIBILITY:
Inclusion Criteria:

* Neonates <28 days of life .
* Hospital stay >48 h .
* Neonates without signs of sepsis at time of admission .
* Accepted to participate in this study .

Exclusion criteria :

* Neonates >28 days of life .
* Hospital stay <48 h .
* Neonates with neonatal sepsis at time of admission.
* Refused to participate in this study .

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates that suspected to have nosocomial infection in neonatal intensive care unit at Assuit University Children hospital
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Bacteriological profile and antibiotic sensitivity of the nosocomial infection in neonatal intensive care unit at Assuit University Children hospital | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Mohamed Mohey, Professor of pediatrics, Principal Investigator — Assiut University; Safwat Mohamed Abdel_Aziz, Assistant professor of pediatr, Principal Investigator — Assiut University

REFERENCES:
- [Background] Fahim NAE. Prevalence and antimicrobial susceptibility profile of multidrug-resistant bacteria among intensive care units patients at Ain Shams University Hospitals in Egypt-a retrospective study. J Egypt Public Health Assoc. 2021 Mar 29;96(1):7. doi: 10.1186/s42506-020-00065-8. PMID 33779849
- [Background] 7. Mahmoud Mohammed GSED, Shoriet AH, Abdel-Aziz SM. Incidence and risk factors of health-care-associated infection in the neonatal intensive care unit of Assiut University Children's Hospital. Journal of Current Medical Research and Practice. 2021;6(1):48-53.
- [Background] 6. Salem GA. Bacterial contamination in neonatal intensive care units in Misurata, Libya: analysis of causative organisms, biofilm formation, and antimicrobial susceptibility. European Journal of Microbiology and Infectious Diseases. 2024;1(2):66-
- [Background] Silva ACBE, Anchieta LM, Rosado V, Ferreira J, Clemente WT, Coelho JS, Mourao PHO, Romanelli RMC. Antimicrobial use for treatment of healthcare-associated infections and bacterial resistance in a reference neonatal unit. J Pediatr (Rio J). 2021 May-Jun;97(3):329-334. doi: 10.1016/j.jped.2020.06.001. Epub 2020 Jun 24. PMID 32592659
- [Background] 4. Koech CC, Rono SJ, Ngeiywa MM, Jeruto P. Neonatal Factors Predisposing Neonates to Nosocomial Infections at Moi Teaching and Referral Hospital. International Journal of Education, Science and Social Sciences. 2024;3(2):35-43.
- [Background] 3. Shwetabh R, Upadhyay MR, Upadhyay R. Aetiological Agents in Neonatal Nosocomial Sepsis and their Sensitivity Pattern from a Tertiary Care Hospital, Odisha, India: A Crosssectional Study. Seizure. 2022;6:6.
- [Background] 2. Moses SS, Kuruvilla TS, Praveen B. Clinicomicrobiological profile of healthcare associated infections in a neonatal intensive care unit and its relation with environmental surveillance. Panacea Journal of Medical Sciences. 2023;13(1):36-41 .
- [Background] 1. Hogeveen M, Heijting I, Jansen S, de Boode W, Hopman J, Overbeek MGD, et al. Nosocomial infections in neonatal care: a scoping review protocol of published surveillance case definitions. 2021.